CLINICAL TRIAL: NCT00711919
Title: Pitavastatin Evaluation of Atherosclerosis Regression by Intensive Cholesterol-Lowering Therapy
Brief Title: Pitavastatin on Carotid Intima-media Thickness
Acronym: PEACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kyoto Prefectural University of Medicine (Other)
Responsible Party: Hiroaki Matsubara, Kyoto Prefectural University of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-255; UMIN000001229
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Hyperlipidemia; Carotid Artery Diseases
MeSH Terms: conditions — Hyperlipidemias; Carotid Artery Diseases | interventions — pitavastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subjects are receiving Pitavastatin, starting at 2 mg, for 12 months. After administration, serum LDL-cholesterol should be kept between 100 and 80 mg/dL by controlling the dose of Pitavastatin or adding other anti-hyperlipidemia agents other than statins.
  Interventions: Drug: Pitavastatin
- 2 (Active Comparator): Subjects are receiving Pitavastatin, starting at 4 mg, for 12 months. After administration, serum LDL-cholesterol should be kept under 80 mg/dL by controlling the dose of Pitavastatin or adding other anti-hyperlipidemia agents other than statins.
  Interventions: Drug: Pitavastatin

INTERVENTIONS:
Drug: Pitavastatin — comparison of different target levels of lipid lowering using Pitavastatin
  Subjects are receiving Pitavastatin, starting at 2 mg, for 12 months.
  Arms: 1
Drug: Pitavastatin — Subjects are receiving Pitavastatin, starting at 4 mg, for 12 months.
  Arms: 2

SUMMARY:
This study is aimed to analyze the effects of aggressive and conventional lipid lowering therapy with Pravastatin on carotid intima-media thickness (IMT) in patients with hyperlipidemia and abnormal thickening of IMT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having hyperlipidemia
* LDL-C at the time of enrollment is no less than 100
* Common carotid IMT is 1.1 mm and over

Exclusion Criteria:

* Received or planned to receive intervention on carotid arteries during the study period
* Overt liver dysfunction (ALT; 100 IU/L and over)
* Overt renal dysfunction (serum creatinine; 2.0 mg/dL and over)
* Receiving Cyclosporin
* Hyperreactive to Pitavastatin
* During pregnancy or lactation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
absolute changes in carotid intima-media thickness from baseline to final visit | 12 months

SECONDARY OUTCOMES:
relative change in carotid intima-media thickness | 12 months
change in LDL-C, HDL-C, TG and RLP-C | 12 months
change in hs-CRP and IL-6 | 12 months
new onset or recurrence of ischemic heart disease, heart failure, stroke and atherosclerosis obliterans | 12 months
sudden death | 12 months
side effects | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Matsubara, MD, PhD, Study Chair — Kyoto Prefectural University of Medicine
Locations (18):
- Japan (18):
  - Ayabe City Hospital, Ayabe, Kyoto
  - Fukuchiyama City Hospital, Fukuchiyama, Kyoto
  - Saiseikai Kyoto Hospital, Kōtari, Kyoto
  - Takeda Hospital, Kyoto, Kyoto
  - Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Kyoto First Red Cross Hospital, Kyoto, Kyoto
  - Tanabe Central Hospital, Kyōtanabe, Kyoto
  - Kumihama Hospital, Kyōtango, Kyoto
  - Maizuru Medical Center, Maizuru, Kyoto
  - Maizuru Kyosai Hospital, Maizuru, Kyoto
  - Nantan General Hospital, Nantan, Kyoto
  - Meiji University of Integrative Medicine Hospital, Nantan, Kyoto
  - Gakken Toshi Hospital, Sugai, Kyoto
  - Uji Hospital, Uji, Kyoto
  - Kyoto Prefectural Yosanoumi Hospital, Yotsutsuji, Kyoto
  - Shiga Hospital, Higashioumi, Shiga
  - Omihachiman Community Medical Center, Ōmihachiman, Shiga
  - Saiseikai Shigaken Hospital, Rittou, Shiga

REFERENCES:
- [Derived] Clezar CN, Flumignan CD, Cassola N, Nakano LC, Trevisani VF, Flumignan RL. Pharmacological interventions for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2023 Aug 4;8(8):CD013573. doi: 10.1002/14651858.CD013573.pub2. PMID 37565307
- [Derived] Ikeda K, Takahashi T, Yamada H, Matsui K, Sawada T, Nakamura T, Matsubara H; (for the PEACE Investigators). Effect of intensive statin therapy on regression of carotid intima-media thickness in patients with subclinical carotid atherosclerosis (a prospective, randomized trial: PEACE (Pitavastatin Evaluation of Atherosclerosis Regression by Intensive Cholesterol-lowering Therapy) study). Eur J Prev Cardiol. 2013 Dec;20(6):1069-79. doi: 10.1177/2047487312451539. Epub 2012 Jun 11. PMID 22689416